CLINICAL TRIAL: NCT05183594
Title: Pilot Phase 2 Study to Evaluate the Efficacy, Safety and Tolerability of TSUPPORT (a Traditional Chinese Medicine) for Adults With Tourette Syndrome
Brief Title: Evaluate the Efficacy, Safety and Tolerability of TSUPPORT for Adults With Tourette Syndrome
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Tasly Pharmaceuticals, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Supportive Care
Other Study IDs: TSupport-US-01
Record Dates: First submitted 2021-12-22; First posted 2022-01-10 (Actual); Last update posted 2022-01-11 (Actual); Status verified 2022-01

CONDITIONS: Tourette Syndrome
Keywords: Tourette Syndrome
MeSH Terms: conditions — Tourette Syndrome

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- TSupport group (Experimental): Subjects will receive TSupport 4 sachets (5 grams/sachet) orally twice daily. Morning dose and evening dose should be administrated at about the same time every day and irrelevant to meals.
  Supportive care duration: 24 weeks.
  Interventions: Dietary Supplement: TSupport (a Traditional Chinese Medicine)

INTERVENTIONS:
Dietary Supplement: TSupport (a Traditional Chinese Medicine) — TSupport is made up of 11 Chinese medicinal herbs.

SUMMARY:
A 28-week single-arm trial to evaluate the efficacy, safety and tolerability of TSupport (a Traditional Chinese Medicine) for adults with Tourette Syndrome.

DETAILED DESCRIPTION:
This study is to evaluate the efficacy, safety and tolerability of TSupport (a Traditional Chinese Medicine) for adults with Tourette Syndrome, which consists of a screening/wash-out period of up to 6 weeks, a 24-week supportive care period and a 4-week follow-up period. During the first 2-week follow-up period, subjects will continue to receive TSupport at half dose.

After informed consent conducted and signed, subjects will receive TSupport orally twice daily. Morning dose and evening dose should be administrated at about the same time every day and irrelevant to meals.

ELIGIBILITY:
Inclusion Criteria:

1. Male or female adult (aged 18-65) with Tourette Syndrome according to Diagnostic and Statistical Manual of Mental Disorders, Fifth Edition (DSM-V).
2. Total Tic Score (TTS) ≥ 20 on the Yale Global Tic Severity Scale (YGTSS) at screening and baseline.
3. In investigator's opinion the presenting tic symptoms cause at least a moderate degree of distress or impairment.
4. On stable psychiatric medication regimen for a minimum of 4 weeks prior to beginning the trial including medications thought to effect tic symptoms.
5. Females of childbearing potential had a negative pregnancy test, must agree to practiced acceptable double-barrier methods of contraception (or abstinence), and were not pregnant or lactating.
6. Willing to participate voluntarily and sign a written informed consent form.
7. In the opinion of the investigator, the subject is considered likely to comply with the study protocol and to have a high probability of completing the study.

Exclusion Criteria:

1. Medical history consistent with another neurologic condition that may have had accompanying abnormal movements (e.g., Huntington's disease, Parkinson's disease, Sydenham's chorea, Wilson's disease, Mental retardation, Traumatic brain injury, Stroke, Restless legs syndrome);
2. History of schizophrenia, bipolar disorder, or other psychotic disorder; intellectual disability or Autism Spectrum Disorder (Level 2 or 3 functioning - requiring substantial social supports or more);
3. Recent change (less than 4 weeks) in medications that have potential effects on tic severity (such as alpha-2 agonists (guanfacine, clonidine or prazosin), SSRIs, clomipramine, naltrexone, lithium, anxiolytics, topiramate, baclofen, VMAT2 inhibitors, ecopipam or compounds containing delta-9 tetrahydrocannabinol (delta-9-THC) or cannabidiol). Medication change is defined to include dose changes or medication discontinuation.
4. Recent change in behavioral treatment for Tourette syndrome or comorbid conditions (i.e. OCD) within the last 4 weeks or initiation of behavioral therapy for tics within the last 12 weeks.
5. Sexually active males or females who would not commit to utilizing 2 of the approved birth control methods or who would not remain abstinent during the trial and for 90 days (males) or 30 days (females) following the last dose of IP
6. Significant psychoactive substance use disorder within the past 3 months; or the urine drug screen was positive for cocaine, opiates, amphetamines, benzodiazepines or marijuana. Subjects prescribed stable medications that cause positive drug tests e.g. benzodiazepines, dronabinol or psychostimulants will be included as long as they do not test positive for substances unexplained by their prescription medication.
7. Significant lab abnormality:

   1. Platelets ≤ 75,000/mm3
   2. Hemoglobin ≤ 9 g/dl
   3. Neutrophils, absolute ≤ 1000/mm3
   4. Aspartate transaminase (AST) > 3×ULN (upper limit of normal)
   5. Alanine aminotransferase (ALT) > 3×ULN
   6. Creatinine ≥ 2 mg/dl
8. History or presence of any clinically important medical condition that, in the judgment of the investigator, is likely to deteriorate, could be detrimental to the subject, or could affect the subject's ability to complete the study.

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 10 (Estimated)
Dates: Start 2022-03 (Estimated); Primary Completion 2024-03 (Estimated); Study Completion 2024-09 (Estimated)

PRIMARY OUTCOMES:
The change from baseline to Week 24 in Yale Global Tic Severity Scale (YGTSS) total tic score (TTS). | Baseline, Week 24
  The Yale Global Tic Severity Scale (YGTSS) is a semi-structured clinical interview for assessing the severity of tics in children and adults. The YGTSS enables evaluations of number, frequency, intensity, complexity, and interference of motor and phonic tics, covering the past week. Each domain is scored on a 6-point scale (range 0-5) with a separate rating for "overall impairment" regarding the subject's daily life and activities. YGTSS-TTS is the sum of the total motor tic score plus the total phonic tic score ranging from 0-50. Higher scores indicate greater severity/worse outcome. The score of TTS on week 24 will be compared to baseline.

SECONDARY OUTCOMES:
The change from baseline to Week 24 in YGTSS tic-related impairment (TRI) scores. | Baseline, Week 24
  The score of TRI on week 24 will be compared to baseline. The YGTSS ranking of impairment (YGTSS-TRI), with a maximum of 50 points, is based on the impact of the tic disorder on areas of self-esteem, family life, social acceptance, and school scores. Higher scores indicate greater severity/worse outcome.
Mean change from baseline to Week 24 in TS-CGI severity and improvement. | Baseline, Week 2, 4, 6, 8, 10, 12, 16, 20 and 24
  The TS-CGI scale is a 7-point Likert scale that allows the clinician to use all available information to assess the impact of tics on the participant's quality of life. Lower scores indicate better quality of life. Mean score was calculated with TSupport group, on week 2, 4, 6, 8, 10, 12, 16, 20 and 24.
Clinical response rate, defined as a ≥ 30% reduction from baseline on TTS at different check points. | Baseline, Week 2, 4, 6, 8, 10, 12, 16, 20 and 24
  Clinical response defined as a ≥ 30% reduction from baseline on TTS at week 2, 4, 6, 8, 10, 12, 16, 20 and 24. The clinical response rate is the proportion of subjects who achieve clinical response.

CONTACTS AND LOCATIONS:
Overall Officials: Michael H Bloch, MD, PhD, Principal Investigator — Yale University
Locations (1):
- Yale Child Study Center, New Haven, Connecticut, United States

IPD SHARING:
Plan to Share IPD: No